CLINICAL TRIAL: NCT05046548
Title: Double-blind, Placebo-controlled, Randomized Study of Tolerability, Safety and Immunogenicity of the Inactivated Whole-virion Concentrated Purified Coronavirus Vaccine, Produced by FSBSI "Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products", on Volunteers at the Age of 18-60 Years
Brief Title: This is a Double-blind, Placebo-controlled, Randomized Study of the Tolerability, Safety and Immunogenicity of an Inactivated Whole Virion Concentrated Purified Vaccine (CoviVac) Against Covid-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VKI-I / II-08/20
Record Dates: First submitted 2021-08-26; First posted 2021-09-16 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Coronavirus Infections; Vaccine
Keywords: COVID-19; Coronavirus infections; Vaccine; SARS-Cov-2; Immunobiological medicine
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Vaccines; Injections, Intramuscular

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine (Experimental): At Stage I:
  Group 1 - 10 volunteers, Vaccine 0.5 ml, 14 days interval, post-vaccination observation period of 28 days.
  At Stage II:
  Group 1 - 140 volunteers,Vaccine0.5 ml, 14 days interval, post-vaccination observation period of 28 days.
  At Stage III:
  Group 3 - 150 volunteers, Vaccine 0.5 ml, 14 days interval, post-vaccination observation for 6 months.
  Interventions: Biological: Vaccine for intramuscular injection
- Placebo (Placebo Comparator): No active ingredient in the placebo
  At Stage I:
  Group 2 - 5 volunteers, Placebo 0.5 ml, 14 days interval, post-vaccination observation period of 28 days.
  At Stage II:
  Group 2 - 45 volunteers, Placebo 0.5 ml, 14 days interval, post-vaccination observation period of 28 days.
  At Stage III:
  Group 4 - 50 volunteers, Placebo 0.5 ml, 14 days interval, post-vaccination observation period of 6 months.
  Interventions: Other: Placebo comparator (without active ingredient) for intramuscular injection

INTERVENTIONS:
Biological: Vaccine for intramuscular injection — Volunteers (10 at the Stage 1; 140 at the Stage 2; 150 at the Stage 3) will receive the vaccine twice spaced 14 days apart, intramuscularly, at a dose of 0.5 ml
  Arms: Vaccine
Other: Placebo comparator (without active ingredient) for intramuscular injection — Volunteers (5 at the Stage 1; 45 at the Stage 2; 50 at the Stage 3) will receive the vaccine twice spaced 14 days apart, intramuscularly, at a dose of 0.5 ml
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo controlled, multi-center clinical trials of the tolerability, safety and immunogenicity of the inactivated whole-virion concentrated purified vaccine against COVID-19, manufactured by FSBSI "Chumakov FSC R&D IBP RAS", on adult volunteers aged 18-60" (Clinical trials, phase I/II). Study purpose is to assess the tolerability, safety and immunogenicity of the inactivated whole-virion concentrated purified coronavirus vaccine sorbed on adult volunteers aged 18-60.

DETAILED DESCRIPTION:
The study is divided into 3 stages. At Stages I and II of the study, a maximum of 300 healthy volunteers aged 18 to 60 years should be screened, of which 200 volunteers meeting the inclusion criteria and not non-inclusion criteria, should be included and randomized to study the tolerability and safety of the vaccine.

Stage I includes 15 men and women:

Group 1 - 10 volunteers who will receive the Vaccine twice with an interval of 14 days intramuscularly in a dose of 0.5 ml with a post-vaccination observation period of 28 days.

Group 2 - 5 volunteers who will receive placebo twice with an interval of 14 days intramuscularly at a dose of 0.5 ml with a post-vaccination observation period of 28 days.

Stage II includes 185 volunteers:

Group 1 - 140 volunteers who will receive the Vaccine twice with an interval of 14 days intramuscularly in a dose of 0.5 ml with a post-vaccination observation period of 28 days.

Group 2 - 45 volunteers who received placebo twice with an interval of 14 days intramuscularly in a dose of 0.5 ml with a post-vaccination observation period of 28 days.

Stage III of the study, a maximum of 300 volunteers should be screened, of which 200 volunteers, meeting the inclusion criteria and not non-inclusion criteria, should be included and randomized to study the safety and immunogenicity of the vaccine.

Group 3 - 150 volunteers who will receive the vaccine twice with an interval of 14 days intramuscularly in a dose of 0.5 ml with a period of post-vaccination observation for 6 months.

Group 4 - 50 volunteers who will receive placebo twice with an interval of 14 days intramuscularly in a dose of 0.5 ml with a post-vaccination observation period of 6 months.

ELIGIBILITY:
Inclusion criteria:

Volunteers must meet the following inclusion criteria:

* Healthy volunteers (men and women) aged 18-60;
* Written informed consent of volunteers to participate in a clinical trial;
* Volunteers who are able to comply with the requirements of the Protocol (i.e. filling out the Self-Observation Diary, come to control visits);
* For women capable of childbearing, a negative pregnancy test and consent to adhere to adequate contraceptive methods (use of contraceptives within six months after the second vaccination). Women should use contraceptive methods that are more than 90% reliable (cervical caps with spermicide, diaphragms with spermicide, condoms, intrauterine devices), or be sterile or postmenopausal.
* For fertile men, consent to adhere to adequate contraceptive methods for six months after the second vaccination. Men and their sexual partners must use contraceptive methods with more than 90% reliability (cervical caps with spermicide, diaphragms with spermicide, condoms, intrauterine devices), or be sterile.

Non-inclusion criteria:

Volunteers cannot be included in the study if any of the following criteria are met:

* Medical staff of clinics and polyclinics;
* A history of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS) or other coronavirus infection (HCoV-229E, HCoV-OC43, HCoV-NL63, HCoV-HKU1);
* History of contacts with confirmed or suspected cases of SARS-CoV-2 infection within 1 month;
* Positive IgM or IgG to SARS-CoV-2, found at screening (for volunteers of Phases I and II);
* Positive PCR test for SARS-CoV-2 at screening;
* Clinically and/or laboratory (according to PCR) confirmed disease with SARS-CoV-2 coronavirus at the current time or in history;
* Serious post-vaccination reaction (temperature above 40 C, hyperemia or edema more than 8 cm in diameter) or complication (collapse or shock-like state that developed within 48 hours after vaccination; convulsions, accompanied or not accompanied by a febrile state) to any previous vaccination in history;
* Aggravated allergic history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, history of serum sickness, history of hypersensitivity or allergic reactions to the administration of any vaccines, known allergic reactions to vaccine components, etc.);
* History of Guillain-Barré syndrome (acute polyradiculitis);
* Previous vaccination with rabies vaccines less than 2 months before immunization or planned vaccination with rabies vaccines within 1 month after immunization with investigational vaccines;
* Vaccination with any other vaccine within 1 month preceding vaccination;
* A history of leukemia, tuberculosis, cancer, autoimmune diseases;
* Positive blood test for HIV, syphilis, hepatitis B/C;
* Volunteers who received immunoglobulin preparations or blood transfusions within the last 3 months prior to the start of the study based on the history;
* Long-term use (more than 14 days) of immunosuppressants or other immunomodulatory drugs during the six months preceding the study, according to the history;
* Any history of any confirmed or suspected immunosuppressive or immunodeficient condition;
* Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, gastrointestinal tract, liver, kidneys, hematopoietic, immune systems, mental illness in exacerbation stage or decompensation stage (recovery earlier than 4 weeks before vaccination) in history;
* Disorder of blood clotting, a tendency to thrombosis in the anamnesis;
* Progressive neurological pathology, a history of convulsive syndrome;
* Diabetes mellitus, hyperthyroidism or other endocrine diseases in history;
* Treatment with glucocorticosteroids, including low doses, as well as topical use of drugs containing steroids (> 10 mg prednisolone, or an equivalent, for more than 14 days in the last three months);
* According to the anamnesis, the volunteer was/is registered in a tuberculosis dispensary and/or a narcological dispensary and/or a neuropsychiatric dispensary and/or others;
* Acute infectious diseases (recovery earlier than 4 weeks before vaccination) according to the history;
* Taking more than 10 units of alcohol per week or anamnestic information about alcoholism, drug addiction, or drug abuse;
* Smoking more than 10 cigarettes a day;
* Participation in any other clinical study within the last 3 months;
* Pregnancy or breastfeeding;
* Axillary temperature at the time of vaccination is more than 37.0 °C;
* Body mass index less than 18 or more than 28 kg/m2;
* Serious concomitant diseases or pathological conditions not listed above, which, according to the investigator, could complicate the evaluation of the study results, including pathological deviations from the age norms and laboratory norms of blood and urine parameters, clinically significant, according to the investigator.

Exclusion criteria:

* Withdrawal of informed consent by a volunteer;
* Serious adverse events or adverse events that do not meet the criteria for severity, the development of which, in the opinion of the investigator, may be detrimental to the health or well-being of the volunteer;
* The need for procedures and/or drug treatment not permitted by the Study Protocol;
* The volunteer was included in violation of the inclusion/non-inclusion criteria of the Protocol;
* The emergence of non-inclusion criteria during the study;
* The need for surgical intervention;
* Any condition in a volunteer requiring, in the reasonable opinion of the investigating physician, the withdrawal of the volunteer from the study;
* The volunteer refuses to cooperate or is undisciplined (for example, not showing up for a planned visit without warning the investigator and/or losing contact with the volunteer), or has dropped out of observation;
* For administrative reasons (termination of the study by the Sponsor or regulatory authorities), as well as for gross violations of the protocol that could affect the study results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2020-10-03 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) | 28 days after second vaccination / placebo
  The percentage of volunteers with an increase in geometric mean titer of specific antibodies (GMT) on day 28 after the second dose of vaccine / placebo in the virus neutralization test and ELISA.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) | 7 and 14 days after the first vaccination / placebo
  Percentage of volunteers with a fourfold (or more) level of seroconversion in the neutralization test and ELISA on days 7 and 14 after the first dose of vaccine / placebo; on day 7, day 14, day 28, 2 months, 3 months, 4 months, 5 months, 6 months after the second dose of vaccine / placebo.
Seroconversion rate [Time frame: 7 and 14 days after first vaccination / placebo] | Percentage of volunteers with a fourfold (or more) level of seroconversion in the neutralization reaction and the ELISA reaction on days 7 and 14 after the first dose of vaccine / placebo; on day 7, day 14, day 28, 2 months, 3 months, 4 months, 5 months,
  Seroconversion rate on day 7, day 14, day 28, 2 months, 3 months, 4 months, 5 months, 6 months after second vaccination / placebo.
Level of γ-IFN and subpopulation composition of T-lymphocytes | 7 and 14 days after the first vaccination / placebo
  Levels of γ-IFN and subpopulation composition of T-lymphocytes on days 7 and 14 after the administration of the first dose of vaccine / placebo; on day 7, day 14, day 28, 2 months, 3 months, 4 months, 5 months, 6 months, after the second dose of vaccine / placebo.
Cases of acute respiratory diseases (influenza, acute respiratory infections, COVID-19) | Within 6 months after the second vaccination / placebo
  The frequency of acute respiratory infections (influenza, acute respiratory infections, COVID-19) within six months after the second dose of vaccine / placebo.
Cases of acute respiratory diseases (influenza, acute respiratory infections, COVID-19) | Within 6 months after the second vaccination / placebo
  The severity of acute respiratory infections (influenza, acute respiratory infections, COVID-19) within six months after the second dose of vaccine / placebo.
Cases of acute respiratory diseases (influenza, acute respiratory infections, COVID-19) | Within 6 months after the second vaccination / placebo
  The duration of acute respiratory infections (influenza, acute respiratory infections, COVID-19) within six months after the second dose of vaccine / placebo.
Frequency and severity of adverse events | Within 6 months after the first dose of vaccine / placebo
  The incidence and severity of adverse events throughout the study period after the first dose of vaccine / placebo
Assessment of adverse events | within 6 months after the first dose of vaccine / placebo
  The incidence of adverse events during the study
Evaluation of clinically significant abnormalities in vital signs | within 6 months after the first dose frame of vaccine / placebo
  The incidence of clinically significant deviations from the main indicators of vital functions.
Evaluation of clinically significant deviations from laboratory parameters | 3, 7, 10 and 14 days after the first vaccination; 4, 7, 14 and 28 days after the second vaccination
  The incidence of clinically significant deviations from the laboratory parameters.
Cases of early termination of participation of volunteers in the study | within 6 months after the introduction of the first dose of vaccine / placebo
  Cases of early termination of the volunteer's use in suggesting the development of AE / SAE associated with the use of study drugs.

CONTACTS AND LOCATIONS:
Locations (5):
- Russia (5):
  - Federal State Budgetary Educational Institution of Higher Education Kirov State Medical University of the Ministry of Health of Russia, Kirov
  - FSBSI Chumakov FSC R&D IBP RAS, Moscow
  - FGBUZ MSCh No. 163 FMBA of Russia, Novosibirsk
  - Eco-Safety Scientific Research Center LLC, Saint Petersburg
  - Center for Family Medicine Joint Stock Company (CSM JSC), Yekaterinburg